CLINICAL TRIAL: NCT04046185
Title: PD-1 Inhibitor Combined With Progesterone Treatment in Early Stage Endometrial Cancer Patients Who Want to Preserve Fertility
Brief Title: Programmed Death-1(PD-1) Inhibitor Combined With Progesterone Treatment in Endometrial Cancer
Acronym: ECCT
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai First Maternity and Infant Hospital (Other)
Responsible Party: Principal Investigator, Xiaoping Wan, Dean, Professor, Shanghai First Maternity and Infant Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ECCT001
Record Dates: First submitted 2019-07-26; First posted 2019-08-06 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Endometrial Cancer Stage I
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Progesterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pd-1 inhibitor and progesterone (Experimental): Toripalimab. 240mg intravenous injection, every 3 weeks, 4 times. Megestrol Acetate Tablets, 160mg, po, once a day.
  Interventions: Drug: PD-1 inhibitor combined progesterone
- progesterone (Active Comparator): Megestrol Acetate Tablets, 160mg, po, once a day.
  Interventions: Drug: progesterone

INTERVENTIONS:
Drug: PD-1 inhibitor combined progesterone — Toripalimab combine with progesterone
  Other Names: Toripalimab combine with progesterone
  Arms: pd-1 inhibitor and progesterone
Drug: progesterone — progesterone
  Arms: progesterone

SUMMARY:
We want to make a comparison of PD-1 inhibitor combined with progesterone versus progesterone alone in the treatment of early stage endometrial cancer patients who want to preserve fertility.

DETAILED DESCRIPTION:
Approximately 63,400 new cases of endometrial cancer are diagnosed annually in China. While the initial treatment for early-stage disease is surgical staging with lymphadenectomy, it is apparently inappropriate for young patients who want to preserve fertility. Currently the standardize treatment for these patients are high-dose progesterone, which will be effective in approximately 40~70% patients. Mirena have been used recently as a new available treatment option, however, no concrete evidence shows it is more effective than the traditional progesterone treatment.

PD-1 inhibitor has been utilized as a salvage treatment in many cancers including ovarian cancer, cervical cancer, lung cancer, gastric cancer and endometrial cancer. As endometrial cancer showed high microsatellite instability-high/deficient mismatch repair (MSI-H/dMMR) rates, it is assumed to be highly responsive to PD-1 inhibitor treatment. Published clinical trial results showed that PD-1 inhibitor treatment was effective in 6/24 late-stage endometrial cancer patients, with little or mild side effects. Here we want to investigate the efficacy of PD-1 inhibitor combined with progesterone in early stage endometrial cancer patients who want to preserve fertility.

ELIGIBILITY:
Inclusion Criteria:

1. Early endometrial cancer patients (cancer confined in the endometrium, endometrioid histology, G1-2)
2. Patients want to preserve fertility
3. Informed consent acquired
4. Age <18, >= 45
5. Eastern Cooperative Oncology Group (ECOG) performance status score <=1
6. Normal blood routine test
7. Normal hepatic and renal function
8. Normal thyroid function
9. Patients willing to accept three times of hysteroscopy: before treatment, 3 months after treatment, 6 months after treatment.
10. Pregnancy test negative before treatment

Exclusion Criteria:

1. Patients are receiving immune-checkpoint inhibitor therapy
2. Patients need or request to receive other anti-cancer drug treatment such as chemotherapy
3. Patients are allergic to immune-checkpoint inhibitor agents
4. Patients have abnormal blood routine test results or impaired hepatic and renal functions
5. Patients have a history of cardiovascular disease, including severe hypertension, frequent cardiac arrhythmia, history of myocardial infarction
6. Patients have a history of hepatitis B or hepatitis C infection, with detectable virus load
7. Severe obstructive lung disease
8. Autoimmune disease
9. Need to receive daily corticosteroid or other immune-inhibitory agents
10. Active tuberculosis patients
11. Patients have a history of other malignant tumors
12. Patients with acute infectious disease

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete remission rate of endometrial curettage tissues | 6 months
  Hysteroscopy was performed 6 months after treatment. If the pathological results are normal, it is considered to be complete remission
Pathologic partial remission rate of endometrial curettage tissues | 6 months
  Hysteroscopy was performed 6 months after treatment. If the pathological results showed hyperplasia, it is considered to be partial remission

SECONDARY OUTCOMES:
adverse effects | up to 1 year after treatment
  side effects was evaluated every 2 weeks during treatment
pregnancy rate | up to 2 years after treatment
  pregnancy rate was recorded after treatment